CLINICAL TRIAL: NCT02410798
Title: Early Feasibility Clinical Study to Investigate the Safety and Performance of TransLoc® Electrodes for Temporary Diaphragm Pacing in Patients Undergoing Surgical Procedures
Brief Title: Clinical Study to Investigate Safety and Performance of TransLoc Electrodes in Patients Undergoing Surgical Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synapse Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN 20-1000-0006
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Diaphragm Pacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TransLoc electrode (Experimental): Electrode placement
  Interventions: Device: TransLoc electrode

INTERVENTIONS:
Device: TransLoc electrode — Patients will have 2 electrodes placed in either side of the diaphragm (total 4 electrodes) during their primary surgery.

SUMMARY:
Feasibility study to advance the development of NeuRx Diaphragm Pacing System (DPS) for the intended use of stimulating the diaphragm to provide respiratory assistance in patients at risk of prolonged mechanical ventilation in the Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
This is a prospective, open-label, single-center study to examine the feasibility of the TransLoc DPS electrode placement and removal. Twelve (12) subjects undergoing a surgical procedure will receive the device (four electrodes) and will be followed until electrode removal up to seven days post-procedure. Subjects will be selected from surgical candidates undergoing laparoscopic, open abdominal, and open thoracic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing a surgical procedure with expected admission to the hospital.
* Patient is undergoing a laparoscopic, open abdominal, or open chest surgical procedure that allows access to the diaphragm.
* Negative pregnancy test if the patient is a female of child-bearing potential.
* Patient is at least 18 years of age.
* Informed consent has been obtained from the patient or designated representative.

Exclusion Criteria:

* Patient has an implanted cardiac defibrillator.
* Patient is pregnant or breastfeeding.
* The patient is involved in another clinical study that could influence the safety or outcome measures of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Onders, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospital, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TransLoc Electrode
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TransLoc Electrode
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 67.6 [41 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant That Experience Adverse Procedure and/or Device Effects
Description: All participants were monitored for adverse device effects (procedure and device related adverse events) from implantation of the TransLoc electrodes through electrode removal.
Time Frame: Implantation through hospital discharge or Day 7, whichever comes first.
Population: Twelve (12) subjects undergoing a surgical procedure will receive the device (four electrodes). Subjects will be selected from surgical candidates undergoing laparoscopic, open abdominal, and open thoracic procedures. Four subjects in each surgical category will be studied.
Measure: Number; unit: Events
Groups:
- Treatment: Patients will have 2 TransLoc electrodes placed in either side of the diaphragm (total 4 electrodes) during their primary surgery.
Arm/Group | Treatment
Number analyzed (Participants) | 12
Events | 0

2. Primary Outcome: Number of Study Participants That Experience Successful Placement of Two Electrodes in Each Hemi-diaphragm
Description: Successful placement of two TransLoc electrodes in each hemi-diaphragm of the study participants during the operative procedure. Success was the ability to perform stimulation postoperatively using the implanted electrodes to effectively stimulate the patients for ventilation as evidenced by the ability to successfully achieve the predicted tidal volume.
Time Frame: Postoperatively on Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 12

3. Primary Outcome: Device Stimulation Using Four Electrodes Will Achieve the Predicted Tidal Volume for Study Participants
Description: Ability of device stimulation using four electrodes to achieve or exceed the percent of predicted tidal volume for all study participant.
Time Frame: Postoperatively Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of predicted tidal volume
Arm/Group | Treatment
Number analyzed (Participants) | 12
Percentage of predicted tidal volume | 137 (30)

4. Primary Outcome: Number of Study Participants in Which Daily Diaphragm EMG Was Successfully Measured.
Description: Ability to use the implanted electrodes to measure diaphragm EMG activity of both hemi-diaphragms for all study participants.
Time Frame: Postop Day 1 through hospital discharge or Day 7, whichever comes first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 12

5. Primary Outcome: Number of Study Participants in Which TransLoc Electrodes Remained in the Diaphragm Until Removed.
Description: Electrode stability was determined by using the electrodes to record tracings of the diaphragm EMG daily for at least a 10 minute period. The tracings were reviewed to determine diaphragm activity including characterization of diaphragm burst activity, breathing patterns and identification of apneic events, if any. The recordings also confirmed electrode stability (non-displacement and electrical integrity) during the period of temporary implantation.
Time Frame: Postop Day 1 through hospital discharge or 7 days, whichever comes first
Population: Four subjects were enrolled into each of the following surgical procedural groups: laparoscopic, open abdominal and open chest.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 12

6. Primary Outcome: Number of Participants That Experienced Complete Removal of Entire TransLoc Electrode
Description: Number of study participants in which TransLoc electrodes were removed intact without device fragmentation or the occurrence of device or procedure related adverse events. Removal was performed by the healthcare provider by pulling electrodes from the percutaneous entry point. This was done in a similar fashion as a temporary cardiac pacing wire with a slow steady pull in a straight non oblique line.
Time Frame: Postop Day 1 through hospital discharge or Day 7, whichever comes first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 12

7. Secondary Outcome: Comparison of Percentage of Predicted Tidal Volumes Measured.
Description: Achieved percent of predicted tidal volume when stimulated using two-electrodes per hemi-diaphragm.
Time Frame: Postop Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of predicted tidal volume
Groups:
- Treatment: Patients will have 2 TransLoc electrodes placed in each hemi-diaphragm (total 4 electrodes) during their primary surgery.
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of predicted tidal volume | 107 (35)

8. Secondary Outcome: Number of Participants That Achieve a Tidal Volume of at Least 6cc/kg of Predicted Body Weight (PBW)
Description: Number of participants in which stimulation successfully achieves acceptable tidal volumes of at least 6cc/kg of predicted body weight (PBW). This predicted tidal volume measurement is based on the NIH NHLBI ARDS Clinical Network (ARDSnet) MV protocol criteria for Acute Respiratory Lung Syndrome (ARDS) protection resulting from the ALVELOI study.
Time Frame: Postop Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 12

9. Secondary Outcome: Number of Participants With Successful Measurement and Characterization of Diaphragm Activity.
Description: Characterization of diaphragm activity including characterization of diaphragm burst activity, breathing patterns and identification of apneic events, if any for each study participant.
Time Frame: Postop Day 1 through hospital discharge or Day 7, whichever comes first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: All participants were monitored for adverse device effects (procedure and device related adverse events) from implantation of the TransLoc electrodes through electrode removal.
Description: Serious device or procedure adverse device effects.
Groups:
- Treatment: Twelve (12) subjects undergoing a surgical procedure will receive the device (four electrodes). Subjects will be selected from surgical candidates undergoing laparoscopic, open abdominal, and open thoracic procedures. Four subjects in each surgical category will be studied.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No